CLINICAL TRIAL: NCT04011605
Title: Microbial Sampling of Carious Dentin
Status: Withdrawn | Type: Observational
Why Stopped: No longer moving forward with study as of May 2022
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Wyatt R. Hume, DDS PhD, Dean, School of Dentistry, University of Utah
Other Study IDs: 00121555
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biological Sample of Carious Dentin — Dental patient volunteers will have either areas of decayed tooth structure or recurrent caries defective fillings removed using conventional, routine procedures, which will include: local anesthesia; tooth isolation using rubber dam; removal of superficial decay, weakened tooth structure or defective filling materials with rotary tooth cutting instruments; and then removal of softened dentin using sterile sharp spoon excavators, by hand. The limit of dentin removal will be determined by the clinician's estimate of tooth hardness, that is, using present conventional and ethical practice.

SUMMARY:
The School of Dentistry is seeking to determine whether viable microorganisms remain within tooth structure after conventional, mechanical removal of areas of tooth decay, prior to placement or replacement of tooth restorations (fillings). The long-term goal of the work is to decrease the failure rate, and therefore increase the longevity, of tooth restorations (fillings) in human patients and populations.

DETAILED DESCRIPTION:
It is proposed that with informed consent, and in a sterile operating environment (controlled, micron level-filtered environmental air flow, in addition to conventional instrument sterilization) dental patient volunteers will have either areas of decayed tooth structure or recurrent caries defective fillings removed using conventional, routine procedures, which will include: local anesthesia; tooth isolation using rubber dam; removal of superficial decay, weakened tooth structure or defective filling materials with rotary tooth cutting instruments; and then removal of softened dentin using sterile sharp spoon excavators, by hand. The limit of dentin removal will be determined by the clinician's estimate of tooth hardness, that is, using present conventional and ethical practice. This last step, removal of tissue guided by estimated hardness, is as described above the universally accepted standard.

Following removal, the exposed dentin surface will be examined visually with an 15X operating microscope to detect any areas of discolored dentin. Any such areas will be micro-sampled using ultra slow-speed, 0.2 mm diameter rotary cutting instruments and removal of resultant dentin flakes with sterile fibers. Each prepared cavity will then be restored using conventional tooth filling materials and techniques.

Immediately after removal each dentin flake will be weighed, placed into bacterial transport medium, then sonicated. The transport medium will be divided in two, and separate samples added to bacterial growth medium under anaerobic and aerobic growth conditions. Any viable microorganisms detected will be identified both by conventional plating techniques using visual identification, and by a commercial laboratory using RNA analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-99, Male or Female, No significant systemic illness

Exclusion Criteria:

* Diabetic, Hypertensive, Pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The School of Dentistry will seek dental patient volunteers to participate in the study if patient meets all inclusion and exclusion criteria and is in need of a Class II filling placement. Flyers will be placed in the reception area of the School of Dentistry clinic. Student dentists will also inform study staff if he/she has a patient who meets the inclusion and exclusion criteria of the study. Study staff will approach the patient to seek informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Detection of viable microorganisms | 1 year from study start date
  Should viable microorganisms be detected within tooth structure after conventional, mechanical removal of decayed areas, future studies into the potential effectiveness of various topical antibacterial agents may well follow.

CONTACTS AND LOCATIONS:
Overall Officials: Wyatt R. Hume, DDS, PhD, Principal Investigator — University of Utah School of Dentistry
Locations (1):
- University of Utah School of Dentistry, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided